CLINICAL TRIAL: NCT01082757
Title: Prevalence of the Mutational Status of KRAS in mCRC in Argentine Patients
Brief Title: Prevalence of the Mutational Status of V-Ki-ras2 Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) in Metastatic Colorectal Cancer (mCRC) in Argentine Patients
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Quimica Argentina S.A.I.C (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR62202-513
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal neoplasms; metastasis; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This observational, prospective, multicentric study is being conducted to record the prevalence of KRAS mutations in the Argentine mCRC population.

DETAILED DESCRIPTION:
This is an observational, prospective, non-interventional, single arm, non-comparative, open label, multi-centric, multi-stage study to record the prevalence of KRAS mutations in the Argentine mCRC population. The study is planned to be conducted in 150 centres (50 in each of 3 stages of four months each, enrolling 500 subjects in each stage). Total of subjects: 1500. Demographic information, complete medical history and tumour history related data will be captured in the first visit and if any information is missing, then only another visit will be scheduled. Data captured will be analysed and presented using statistical tools.

OBJECTIVES:

Primary objective:

* To record the prevalence of KRAS mutations in the Argentine mCRC population.

Secondary objective:

* To record and evaluate certain subject and tumour characteristics for association with KRAS mutational status (country, gender, age, performance status, body mass index (BMI), ethnic origin, personal and family history of malignancy, personal and family history of familial polyposis coli, smoking status, exercise, diet, tumour characteristics/location, site of origin of the tissue sample sent for KRAS testing, first line therapy chosen).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have signed written informed consent before any study-related procedure
* Subjects with histologically confirmed adenocarcinoma of the colon/ rectum, T1-4 N0-2 M1 or rT1-4 N0-2 M1
* Subjects with age above 21 years
* Subjects willing to provide information required by protocol
* No previous systemic treatment for mCRC

Exclusion Criteria:

* Subjects with known pregnancy
* Subjects with previous systemic therapy for mCRC
* Subjects with active infection or any other serious condition which, in the investigator´s mind, may render the subject ineligible for the study
* Subjects with medical or psychological condition, which, in the opinion of the investigator, would not permit the subject to sign meaningful informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with histologicaly confirmed metastatic adenocarcinoma of the colon/rectum in Argentina
Sampling Method: Non-Probability Sample
Enrollment: 1524 (Actual)
Dates: Start 2009-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mutational status of KRAS: study of codons 12 and 13 in exon 1 of KRAS gene | Initial visit (Day 1) and subsequent visit till the end of the study

SECONDARY OUTCOMES:
Subject and tumour characteristics and their association with KRAS mutational status | Initial visit (Day 1) and subsequent visit till the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Quimica Argentina S.A.I.C
Locations (1):
- Htal Vicente Lopez, Vicente López, Argentina